CLINICAL TRIAL: NCT05639855
Title: Study on Mental Health-related Stigma: Attitudes and Values of University Students Towards People With Mental Disorders
Brief Title: Study on Mental Health-related Stigma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nereida Canosa Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Nereida Canosa Rodríguez, Professor, Universidade da Coruña
Organization: Universidade da Coruña (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2021/028
Record Dates: First submitted 2022-11-13; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Mental Health Disorder
Keywords: mental health disorder; stigma; university students; occupational therapy; alphabetisation
MeSH Terms: conditions — Mental Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Third year students of the Bachelor's Degree in Occupational Therapy (Experimental): Third-year students of the Bachelor's Degree in Occupational Therapy will receive training on a specific module on mental health and stigma in the university curriculum.
  Interventions: Other: Mental Health Literacy Programme
- Students of University of A Coruña (No Intervention): The students of the University of A Coruña will take part in an online survey to find out the attitudes and beliefs of future professionals from different areas of knowledge regarding mental health.
- People with mental health disorder (No Intervention): Users of a Psychosocial and Labor Rehabilitation Centers in the A Coruña Health Care Area will take part in interviews to find out their experiences regarding the attributions made towards them by citizens and health professionals.

INTERVENTIONS:
Other: Mental Health Literacy Programme — Mental Health Literacy Program. This program is part of the training of third-year students of the occupational therapy degree at the University of A Coruña. We will follow a mixed method following a sequential explanatory design. The quantitative part corresponds to a quasi-experimental study, where a comparison will be made between the phase before and after the students take the program. The qualitative part will comprise a phenomenological study to collect the knowledge acquired by the students after taking the program.
  Arms: Third year students of the Bachelor's Degree in Occupational Therapy

SUMMARY:
Mental disorders are currently among the main causes of disability worldwide. For this reason, various national and international organisations include the promotion of mental health among their strategic actions, with special emphasis on the fight against stigma. Evidence shows that stigma has a negative impact on the process of recovery and participation of people with mental disorders.

The general aim of this study is to find out about the attitudes of university students at the University of A Coruña towards people with mental disorders and specifically to intervene with students of the Bachelor's Degree in Occupational Therapy to assess whether taking part in a Mental Health Literacy Programme changes these attitudes.

DETAILED DESCRIPTION:
In recent years, there has been a growing interest in developing and evaluating anti-stigma plans in the field of mental health. However, stigmatising, coercive or paternalistic attitudes persist in society and have a negative impact on the recovery process of people with mental illness.

The Mental Health Spain Confederation proposes tackling stigma through intersectional mental health literacy interventions that incorporate the gender perspective and are focused on the needs identified by people with mental disorders.

The New Mental Health Strategy of the National Health System (2021-2026) establishes the need to involve people and their families, as well as the different social agents in the fight against stigma, especially social and health professionals, as well as the media and educational personnel. The aim of this study is to understand the nature of stigma towards people with mental disorders. In order to do so, it is necessary to take into consideration the experiences and experiences of the people themselves in order to develop plans to promote mental health from a participatory and comprehensive perspective. Likewise, it is considered relevant to know the perceptions of future professionals from different areas of knowledge (students of the University of A Coruña), evaluating their attitudes and beliefs regarding mental health. Finally, the aim is to evaluate the impact of incorporating a specific module on mental health and stigmatisation. a specific module on mental health and stigma in the university curriculum of the students of the Occupational Therapy Degree.

This research has the following objectives: (1) find out the perception of people with mental disorders in relation to the social stigma of citizens and Health Science professionals; (2) find out how university students perceive people with mental health problems, and (3) evaluate the impact of incorporating a specific module on mental health and stigma in the university curriculum, specifically in the Bachelor's Degree in Occupational Therapy.

ELIGIBILITY:
Inclusion Criteria Group I:

* Be graduated at Occupational Therapy Degree at the University of A Coruña

Exclusion Criteria Group I:

* Have difficulties in understanding and/or communication
* Not being enrolled in the Mental Health module of the Degree in Occupational Therapy

Inclusion Criteria Group II:

* Student in the University of A Coruña

Exclusion Criteria Group II:

* Have difficulties in understanding and/or communication

Inclusion Criteria Group III:

* Have a mental disorder [according to the Diagnostic Manual Diagnostic Manual]
* Be a user of the Psychosocial and Labor Rehabilitation Centers of the Health Area of A Coruña

Exclusion Criteria Group III:

* Have difficulties in understanding and/or communication
* Be in a situation of legal incapacity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes on the measurement of the students of third-year of occupational therapy bachelor's degree attitudes and beliefs toward people with mental disorders | One month pre-intervention and one month post-intervention
  It is composed of 40 items, rated on a 5-point Likert scale, ranging from strongly agree to strongly disagree. The scale comprises 4 factors: authoritarianism, benevolence, social restraint, and mental health ideology in the community. Each factor contains 10 statements concerning opinions about the way people with mental disorder are treated. Five of the 10 items are expressed in the positive and the other 5 are worded in the negative. The score for each subscale results from adding the positive items together with the negative items, which are transformed into positive values, with the total score being the sum of all of them. The higher the score, the greater the agreement. The sum of each factor is analyzed with the mean and standard deviation.
Changes on the measurement of stigmatizing attitudes towards people with mental health disorders in students of third-year of occupational therapy bachelor's degree | One month pre-intervention and one month post-intervention
  It is a Likert-type scale with 27 items on the situation posed, grouped into 9 factors: responsibility, pity, anger, dangerousness, fear, help, coercion, segregation and avoidance. I sum the items of each factor, obtaining a minimum of 3 and a maximum of 27.
Acquired knowledge in students of third-year of occupational therapy bachelor's degree who participated in the intervention programme | within 1 month after the intervention
  The interview is the most used data collection technique in qualitative studies. In this study, a semi-structured interview will be used because it is flexible and dynamic. It's a beginning interview to know the knowledge acquired by the students.

SECONDARY OUTCOMES:
Measurement of the Students of University of A Coruña attitudes and beliefs toward people with mental disorders | within 1 month after the intervention
  It is composed of 40 items, rated on a 5-point Likert scale, ranging from strongly agree to strongly disagree. The scale comprises 4 factors: authoritarianism, benevolence, social restraint and mental health ideology in the community. Each factor contains 10 statements concerning opinions about the way people with mental disorder are treated. Five of the 10 items are expressed in the positive and the other 5 are worded in the negative. The score for each subscale results from adding the positive items together with the negative items, which are transformed into positive values, with the total score being the sum of all of them.
Measurement of stigmatizing attitudes towards people with mental health disorders of the Students of University of A Coruña | within 1 month after the intervention
  It is a Likert-type scale with 27 items on the situation posed, grouped into 9 factors: responsibility, pity, anger, dangerousness, fear, help, coercion, segregation and avoidance. I sum the items of each factor, obtaining a minimum of 3 and a maximum of 27.
Individual-interviews | within 1 month after the intervention
  The interviews were about the experiences of people with mental disorders in relation to stigma. The following questions composed the interview: the definition of stigma, the influence of society on people with a mental health disorder, experiences about the barriers detected in daily life, and the behavior of the health providers that work with people with a mental health disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Nereida Canosa Domínguez, Master, Principal Investigator — Universidade da Coruña
Locations (1):
- Nereida Canosa Domínguez, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan contains the collection of the variables of the present study.

REFERENCES:
- [Result] Hankir AK, Northall A, Zaman R. Stigma and mental health challenges in medical students. BMJ Case Rep. 2014 Sep 2;2014:bcr2014205226. doi: 10.1136/bcr-2014-205226. PMID 25183806
- [Result] Clement S, Schauman O, Graham T, Maggioni F, Evans-Lacko S, Bezborodovs N, Morgan C, Rusch N, Brown JS, Thornicroft G. What is the impact of mental health-related stigma on help-seeking? A systematic review of quantitative and qualitative studies. Psychol Med. 2015 Jan;45(1):11-27. doi: 10.1017/S0033291714000129. Epub 2014 Feb 26. PMID 24569086
- [Result] Corrigan PW, Mittal D, Reaves CM, Haynes TF, Han X, Morris S, Sullivan G. Mental health stigma and primary health care decisions. Psychiatry Res. 2014 Aug 15;218(1-2):35-8. doi: 10.1016/j.psychres.2014.04.028. Epub 2014 Apr 18. PMID 24774076
- [Result] Lanfredi M, Macis A, Ferrari C, Rillosi L, Ughi EC, Fanetti A, Younis N, Cadei L, Gallizioli C, Uggeri G, Rossi R. Effects of education and social contact on mental health-related stigma among high-school students. Psychiatry Res. 2019 Nov;281:112581. doi: 10.1016/j.psychres.2019.112581. Epub 2019 Sep 27. PMID 31586833
- [Result] Mejia-Lancheros C, Lachaud J, O'Campo P, Wiens K, Nisenbaum R, Wang R, Hwang SW, Stergiopoulos V. Trajectories and mental health-related predictors of perceived discrimination and stigma among homeless adults with mental illness. PLoS One. 2020 Feb 27;15(2):e0229385. doi: 10.1371/journal.pone.0229385. eCollection 2020. PMID 32106225
- [Result] Milin R, Kutcher S, Lewis SP, Walker S, Wei Y, Ferrill N, Armstrong MA. Impact of a Mental Health Curriculum on Knowledge and Stigma Among High School Students: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2016 May;55(5):383-391.e1. doi: 10.1016/j.jaac.2016.02.018. Epub 2016 Mar 8. PMID 27126852
- [Result] Mahmoudi H, Saffari M, Movahedi M, Sanaeinasab H, Rashidi-Jahan H, Pourgholami M, Poorebrahim A, Barshan J, Ghiami M, Khoshmanesh S, Potenza MN, Lin CY, Pakpour AH. A mediating role for mental health in associations between COVID-19-related self-stigma, PTSD, quality of life, and insomnia among patients recovered from COVID-19. Brain Behav. 2021 May;11(5):e02138. doi: 10.1002/brb3.2138. Epub 2021 Apr 3. PMID 33811451
- [Result] Adu J, Oudshoorn A, Anderson K, Marshall CA, Stuart H, Stanley M. Policies and Interventions to Reduce Familial Mental Illness Stigma: A Scoping Review of Empirical Literature. Issues Ment Health Nurs. 2021 Dec;42(12):1123-1137. doi: 10.1080/01612840.2021.1936710. Epub 2021 Jul 28. PMID 34319817
- [Result] Ma HI, Hsieh CE. An Anti-Stigma Course for Occupational Therapy Students in Taiwan: Development and Pilot Testing. Int J Environ Res Public Health. 2020 Aug 3;17(15):5599. doi: 10.3390/ijerph17155599. PMID 32756448
- [Result] Tomar N, Ghezzi MA, Brinkley-Rubinstein L, Wilson AB, Van Deinse TB, Burgin S, Cuddeback GS. Statewide mental health training for probation officers: improving knowledge and decreasing stigma. Health Justice. 2017 Nov 15;5(1):11. doi: 10.1186/s40352-017-0057-y. PMID 29143153